CLINICAL TRIAL: NCT02896998
Title: Routine Versus on Demand Removal of the Syndesmotic Screw
Acronym: RODEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.C. Goslings, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METC2016_197
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Anke Fracture; Syndesmotic Injury
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control group (Other): The syndesmotic screw will routinely be removed 8 - 12 weeks following placement of the screw
  Interventions: Procedure: Routine removal of fhe syndesmotic screw
- Intervention (Experimental): The syndesmotic screw will only be removed in case of symptomatic implants (e.g. implants causing pain or restricted range of motion)
  Interventions: Procedure: Removal on demand of the syndesmotic screw

INTERVENTIONS:
Procedure: Removal on demand of the syndesmotic screw — The syndesmotic screw will only be removed in case of a symptomatic implant (e.g. implant causing pain or restricted range of motion)
  Arms: Intervention
Procedure: Routine removal of fhe syndesmotic screw — The syndesmotic screw will routinely be removed 8 - 12 weeks following placement of the screw
  Arms: Control group

SUMMARY:
The objective of this trial is to demonstrate that the functional outcome of 'removal on demand' of the syndesmotic screw is non-inferior compared to routine removal of the syndesmotic screw in patients with an ankle fracture.

ELIGIBILITY:
Inclusion Criteria:

* Over 17 years of age
* Placement of a metallic syndesmotic screw for an unstable ankle fracture or an isolated syndesmotic injury
* Syndesmotic screw placed within two weeks of the trauma
* Being in such condition that one is able to possibly undergo a second procedure

Exclusion Criteria:

* ISS score >15
* Injuries to the ipsi- and contralateral side which might hamper rehabilitation
* Other medical conditions which hamper physical rehabilitation
* Incomprehensive understanding of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2017-01; Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Functional outcome through the Olerud-Moland score | 1 year following initial treatment

SECONDARY OUTCOMES:
Functional outcome through the OAFAS | 1 year following initial treatment
Pain through the Visual Analog scale | 1 year following initial treatment
Range of motion | 1 year following initial treatment
Surgical complications | 1 year following initial treatment
Quality of Life through the EQ-5D-5L | 1 year following initial treatment
Health care consumption through the iMCQ | 1 year following initial treatment
Loss of productivity through the iPCQ | 1 year following initial treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Dingemans SA, Birnie MFN, Sanders FRK, van den Bekerom MPJ, Backes M, van Beeck E, Bloemers FW, van Dijkman B, Flikweert E, Haverkamp D, Holtslag HR, Hoogendoorn JM, Joosse P, Parkkinen M, Roukema G, Sosef N, Twigt BA, van Veen RN, van der Veen AH, Vermeulen J, Winkelhagen J, van der Zwaard BC, van Dieren S, Goslings JC, Schepers T. Routine versus on demand removal of the syndesmotic screw; a protocol for an international randomised controlled trial (RODEO-trial). BMC Musculoskelet Disord. 2018 Jan 31;19(1):35. doi: 10.1186/s12891-018-1946-5. PMID 29386053